CLINICAL TRIAL: NCT01037218
Title: Randomized, Placebo-controlled, Double-Blind, Parallel Design, Phase 3 Study to Assess the Safety and Efficacy of Udenafil Tablets in Male Subjects With Erectile Dysfunction
Brief Title: Treatment of Erectile Dysfunction II
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Warner Chilcott (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PR-01309
Record Dates: First submitted 2009-10-19; First posted 2009-12-22 (Estimated); Results first posted 2011-12-22 (Estimated); Last update posted 2015-06-19 (Estimated); Status verified 2015-05

CONDITIONS: Erectile Dysfunction
MeSH Terms: conditions — Erectile Dysfunction | interventions — udenafil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Udenafil 50 mg (Experimental): 50 mg Udenafil tablet plus 100 & 150 mg placebo tablets
  Interventions: Drug: Udenafil; Drug: Placebo
- Udenafil 100 mg (Experimental): 100 mg Udenafil tablet plus 50 & 150 mg placebo tablets
  Interventions: Drug: Udenafil; Drug: Placebo
- Udenafil 150mg (Experimental): 150 mg Udenafil tablet plus 50 & 100 mg placebo tablets
  Interventions: Drug: Udenafil; Drug: Placebo
- Placebo (Placebo Comparator): 50, 100 & 150 mg placebo tablets
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Udenafil — Tablets via oral administration before an attempt at sexual intercourse.
  Arms: Udenafil 100 mg; Udenafil 150mg; Udenafil 50 mg
Drug: Placebo — Tablets via oral administration before an attempt at sexual intercourse.

SUMMARY:
Randomized, placebo-controlled, double-blind, parallel design, Phase 3 study to evaluate the safety and efficacy of udenafil, an orally administered, potent and selective inhibitor of PDE-5 versus placebo for the treatment of subjects with erectile dysfunction (ED).

DETAILED DESCRIPTION:
Multi-center, randomized, double-blind, placebo-controlled, parallel-group design, Phase 3 pivotal study to investigate the efficacay and safety of 50 mg, 100 mg and 150 mg udenafil tablets compared with placebo in men with ED. This study consisted of a 4-week, treatment free run-in period followed by a treatment period of 12 weeks, with an on-demand dosing regimen.

ELIGIBILITY:
Inclusion Criteria:

* Male, at least 19 years of age
* Stable monogamous relationship for at least 6 months with a consenting female partner who is at least 19 years of age, vaginal intercourse is a required study activity
* History of ED (clinically defined as the inability to attain and maintain an erection of the penis sufficient to permit satisfactory sexual intercourse) of at least 3 months duration
* Partner is not pregnant or lactating

Exclusion Criteria:

* History of new-onset symptomatic coronary artery disease within the last 3 months or a history of myocardial infarction or cardiac surgical procedure within six months
* Cardiac arrhythmias requiring antiarrhythmic treatment
* Symptomatic congestive heart failure
* Taking nitrate medication in any form
* Uncontrolled diabetes (HbA1c ≥ 13%)
* Hypersensitivity to phosphodiesterase type 5 (PDE-5) inhibitors such as Viagra®, Cialis® or Levitra®
* Previously failed to respond to PDE-5 inhibitors such as Viagra®, Cialis® or Levitra®

Min Age: 19 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 601 (Actual)
Dates: Start 2009-09; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Herman Ellman, MD, Study Director — Warner Chilcott
Locations (39):
- United States (39):
  - Warner Chilcott Investigational Site, Birmingham, Alabama
  - Warner Chilcott Investigational Site, Huntsville, Alabama
  - Warner Chilcott Investigational Site, Tempe, Arizona
  - Warner Chilcott Investigational Site, Chino, California
  - Warner Chilcott Investigational Site, Tarzana, California
  - Warner Chilcott Investigational Site, Englewood, Colorado
  - Warner Chilcott Investigational Site, Milford, Connecticut
  - Warner Chilcott Investigational Site, Aventura, Florida
  - Warner Chilcott Investigational Site, Daytona Beach, Florida
  - Warner Chilcott Investigational Site, DeLand, Florida
  - Warner Chilcott Investigational Site, Ocala, Florida
  - Warner Chilcott Investigational Site, Tampa, Florida
  - Warner Chilcott Investigational Site, Dawsonville, Georgia
  - Warner Chilcott Investigational Site, Sandy Springs, Georgia
  - Warner Chilcott Investigational Site, Fort Wayne, Indiana
  - Warner Chilcott Investigational Site, Greenwood, Indiana
  - Warner Chilcott Investigational Site, West Des Moines, Iowa
  - Warner Chilcott Investigational Site, Elkridge, Maryland
  - Warner Chilcott Investigational Site, Greenbelt, Maryland
  - Warner Chilcott Investigational Site, Las Vegas, Nevada
  - Warner Chilcott Investigational Site, Lawrenceville, New Jersey
  - Warner Chilcott Investigational Site, Bay Shore, New York
  - Warner Chilcott Investigational Site, Brooklyn, New York
  - Warner Chilcott Investigational Site, Kingston, New York
  - Warner Chilcott Investigational Site, New York, New York
  - Warner Chilcott Investigational Site, Poughkeepsie, New York
  - Warner Chilcott Investigational Site, Williamsville, New York
  - Warner Chilcott Investigational Site, Cary, North Carolina
  - Warner Chilcott Investigational Site, Raleigh, North Carolina
  - Warner Chilcott Investigational Site, Salisbury, North Carolina
  - Warner Chilcott Investigational Site, Cleveland, Ohio
  - Warner Chilcott Investigational Site, Jenkintown, Pennsylvania
  - Warner Chilcott Investigational Site, Lancaster, Pennsylvania
  - Warner Chilcott Investigational Site, Greer, South Carolina
  - Warner Chilcott Investigational Site, Arlington, Texas
  - Warner Chilcott Investigational Site, San Antonio, Texas
  - Warner Chilcott Investigational Site, Norfolk, Virginia
  - Warner Chilcott Investigational Site, Richmond, Virginia
  - Warner Chilcott Investigational Site, Mountlake Terrace, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First Subject enrolled 28-Sep-2009
Groups:
- Udenafil 50 mg: Udenafil 50 mg tablets
- Udenafil 100 mg: Udenafil 100 mg tablets
- Udenafil 150mg: Udenafil 150mg tablets
- Placebo: Placebo tablets
Period: Overall Study
Arm/Group | Udenafil 50 mg | Udenafil 100 mg | Udenafil 150mg | Placebo
Started | 147 | 149 | 155 | 150
Safety Population | 147 | 148 | 154 | 150
mITT Population | 141 | 140 | 147 | 141
Completed | 131 | 128 | 134 | 134
Not Completed | 16 | 21 | 21 | 16
Not completed — Adverse Event | 4 | 2 | 2 | 1
Not completed — Lack of Efficacy | 0 | 2 | 1 | 5
Not completed — Lost to Follow-up | 3 | 5 | 4 | 2
Not completed — Withdrawal by Subject | 6 | 7 | 7 | 4
Not completed — Partner Withdrew Consent | 0 | 3 | 2 | 1
Not completed — Protocol Violation | 0 | 0 | 2 | 2
Not completed — Various | 3 | 2 | 3 | 1

BASELINE CHARACTERISTICS:
Population: Subjects Randomized/Enrolled; Age, Ethnic, Race only available for Safety Population
Groups:
- Total: Total of all reporting groups
Arm/Group | Udenafil 50 mg | Udenafil 100 mg | Udenafil 150mg | Placebo | Total
Number analyzed (Participants) | 147 | 149 | 155 | 150 | 601
Age, Continuous [Mean (Standard Deviation); unit: years] — Safety Population
  years | 59.1 (8.92) | 56.8 (10.22) | 58.7 (9.48) | 58.9 (10.31) | 58.4 (9.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 147 | 149 | 155 | 150 | 601
Ethnicity (NIH/OMB) [Number; unit: Participants] — Race Safety Population
  Participants
    Hispanic or Latino | 7 | 5 | 9 | 8 | 29
    Not Hispanic or Latino | 140 | 143 | 145 | 142 | 570
    Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Number; unit: Participants] — Safety Population
  Participants
    American Indian or Alaska Native | 1 | 2 | 1 | 0 | 4
    Asian | 0 | 1 | 1 | 1 | 3
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
    Black or African American | 17 | 20 | 13 | 19 | 69
    White | 129 | 125 | 139 | 127 | 520
    More than one race | 0 | 0 | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0 | 3 | 3
Region of Enrollment [Number; unit: participants]
  United States | 147 | 149 | 155 | 150 | 601

OUTCOME MEASURES:

1. Primary Outcome: Change in Erectile Function Domain Assessed by International Index of Erectile Function (IIEF), Baseline to Final Visit/Week 12, mITT (Modified Intent-to-Treat), LOCF (Last Observation Carried Forward)
Description: Erectile Function domain: 0 - 5 scoring scale for each of 6 questions (scale: 0/min/poor - 30/max/good). Over last month: How often were you able to get erection? When you had erections with stimulation, how often were your erections hard enough for penetration? When you attempted intercourse, how often were you able to penetrate your partner? How often were you able to maintain your erection after penetrating your partner? How difficult was it to maintain your erection to completion of intercourse? How do you rate your confidence that you can get & keep your erection?
Time Frame: Baseline and Week 12
Population: mITT, LOCF
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a Scale
Arm/Group | Udenafil 50 mg | Udenafil 100 mg | Udenafil 150mg | Placebo
Number analyzed (Participants) | 141 | 140 | 147 | 141
Units on a Scale | 3.79 [2.58 to 5.00] | 6.14 [4.92 to 7.37] | 7.94 [6.75 to 9.12] | 0.41 [-0.81 to 1.62]
Statistical Analysis 1: Comparison: Udenafil 50 mg vs Placebo; 540 subjects were randomized with 1:1:1:1 randomization scheme to the 4 treatment groups (placebo and udenafil 50mg, 100mg or 150mg). 135 subjects for each group vs. Placebo will provide at least 90% power with effect size from 0.41-0.44, 0.74-0.90 and 0.46-0.95 on 50 mg, 100 mg and 150 mg groups, respectively. Adjusted power is at least 90% using Bonferroni adjustment on hierarchical testing procedure. Considerations are based on results from Phase 2, Dong-A Study DA 2005-001 (NCT00282607); Test type: Superiority or Other; p < 0.0001, ANCOVA; Baseline domain score and pooled site as covariates; Difference in LS Means = 3.38, 95% CI 2-sided [1.70 to 5.07]
Statistical Analysis 2: Comparison: Udenafil 100 mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA; Baseline domain score and pooled site as covariates; Difference in LS Means = 5.74, 95% CI 2-sided [4.05 to 7.43]
Statistical Analysis 3: Comparison: Udenafil 150mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA; Baseline domain score and pooled site as covariates; Difference in LS Means = 7.53, 95% CI 2-sided [5.86 to 9.20]

2. Primary Outcome: Changes in Sexual Encounter Profile (SEP), Question 2, Change From Baseline to Overall Study/Weeks 1-12, mITT
Description: Question 2 SEP: Were you able to insert your penis into your partner's vagina? yes/no response. Percent yes responses at baseline compared with percent yes responses in overall study treatment period.
Time Frame: Baseline and Weeks 1-12
Population: mITT
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage of Yes Reponses
Arm/Group | Udenafil 50 mg | Udenafil 100 mg | Udenafil 150mg | Placebo
Number analyzed (Participants) | 141 | 140 | 147 | 141
Percentage of Yes Reponses | 14.47 [9.60 to 19.33] | 19.34 [14.46 to 24.23] | 27.12 [22.39 to 31.85] | -5.72 [-10.57 to -0.86]
Statistical Analysis 1: Comparison: Udenafil 50 mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA; P-values were obtained from ANCOVA model with proportion of "yes" responses during the baseline period and pooled site as covariates; Difference in LS Means = 20.19, 95% CI 2-sided [13.44 to 26.93]
Statistical Analysis 2: Comparison: Udenafil 100 mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 2, analysis 1]; Difference in LS Means = 25.06, 95% CI 2-sided [18.32 to 31.81]
Statistical Analysis 3: Comparison: Udenafil 150mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 2, analysis 1]; Difference in LS Means = 32.84, 95% CI 2-sided [26.18 to 39.50]

3. Primary Outcome: Changes in Sexual Encounter Profile (SEP), Question 3, Change From Baseline to Overall Study/Weeks 1-12, mITT
Description: Question 3 SEP: Did your erection last long enough for you to have successful completion of intercourse? yes/no response. Percent yes responses at baseline compared with percent yes responses in overall study treatment period.
Time Frame: Baseline and Weeks 1-12
Population: mITT
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage of Yes Responses
Arm/Group | Udenafil 50 mg | Udenafil 100 mg | Udenafil 150mg | Placebo
Number analyzed (Participants) | 141 | 140 | 147 | 141
Percentage of Yes Responses | 33.24 [27.81 to 38.67] | 38.34 [32.89 to 43.80] | 46.93 [41.66 to 52.20] | 11.53 [6.10 to 16.95]
Statistical Analysis 1: Comparison: Udenafil 50 mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 2, analysis 1]; Difference in LS Means = 21.72, 95% CI 2-sided [14.19 to 29.24]
Statistical Analysis 2: Comparison: Udenafil 100 mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 2, analysis 1]; Difference in LS Means = 26.82, 95% CI 2-sided [19.27 to 34.37]
Statistical Analysis 3: Comparison: Udenafil 150mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 2, analysis 1]; Difference in LS Means = 35.41, 95% CI 2-sided [27.98 to 42.83]

4. Secondary Outcome: Change in Satisfaction of Intercourse Domain Score Assessed by IIEF, Baseline to Week 12/Final Visit, mITT, LOCF
Description: Satisfaction of Intercourse domain: 0 (poor) - 5/(good) scoring scale for each of 3 questions (0-15/good). Over last month: How many times have you attempted sexual intercourse? When you attempted intercourse, how often was it satisfactory for you? How much have you enjoyed sexual intercourse?
Time Frame: Baseline and Week 12
Population: mITT, LOCF
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a Scale
Arm/Group | Udenafil 50 mg | Udenafil 100 mg | Udenafil 150mg | Placebo
Number analyzed (Participants) | 141 | 140 | 147 | 141
Units on a Scale | 1.49 [0.97 to 2.00] | 2.25 [1.73 to 2.76] | 2.86 [2.36 to 3.36] | -0.04 [-0.55 to 0.47]
Statistical Analysis 1: Comparison: Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA; P-values are obtained from ANCOVA model with Baseline domain score and pooled site as covariates; Difference in LS Means = 1.52, 95% CI 2-sided [0.81 to 2.23]
Statistical Analysis 2: Comparison: Udenafil 100 mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA; P-values are obtained from ANCOVA model with Baseline domain score and pooled site as covariates; Difference in LS Means = 2.29, 95% CI 2-sided [1.58 to 3.00]
Statistical Analysis 3: Comparison: Udenafil 150mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA; P-values are obtained from ANCOVA model with Baseline domain score and pooled site as covariates; Difference in LS Means = 2.90, 95% CI 2-sided [2.20 to 3.60]

5. Secondary Outcome: Change in Orgasmic Function Domain Score Assessed by IIEF, Baseline to Week 12/Final Visit, mITT, LOCF
Description: Orgasmic Function domain: 0/poor - 5/good scoring scale for each of 2 questions (0-10/good). Over last month, when you had sexual stimulation or intercourse how often did you ejaculate? When you had sexual stimulation or intercourse how often did you have the feeling of orgasm (with or without ejaculation)?
Time Frame: Baseline and Week 12
Population: mITT, LOCF
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a Scale
Arm/Group | Udenafil 50 mg | Udenafil 100 mg | Udenafil 150mg | Placebo
Number analyzed (Participants) | 141 | 140 | 147 | 141
Units on a Scale | 0.84 [0.38 to 1.29] | 1.77 [1.32 to 2.23] | 1.78 [1.33 to 2.22] | 0.25 [-0.21 to 0.70]
Statistical Analysis 1: Comparison: Udenafil 50 mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0673, ANCOVA; P-values are obtained from ANCOVA model with Baseline domain score and pooled site as covariates; Difference in LS Means = 0.59, 95% CI 2-sided [-0.04 to 1.22]
Statistical Analysis 2: Comparison: Udenafil 100 mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA; P-values are obtained from ANCOVA model with Baseline domain score and pooled site as covariates; Difference in LS Means = 1.53, 95% CI 2-sided [0.90 to 2.16]
Statistical Analysis 3: Comparison: Udenafil 150mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA; P-values are obtained from ANCOVA model with Baseline domain score and pooled site as covariates; Difference in LS Means = 1.53, 95% CI 2-sided [0.91 to 2.15]

6. Secondary Outcome: Change in Sexual Desire Domain Score Assessed by IIEF, Baseline to Week 12/Final Visit, mITT, LOCF
Description: Sexual Desire domain: 1/poor - 5/good scoring scale for each of 2 questions (2-10/good). Over last month, how often have you felt sexual desire? How would you rate your level of sexual desire?
Time Frame: Baseline and Week 12
Population: mITT, LOCF
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a Scale
Arm/Group | Udenafil 50 mg | Udenafil 100 mg | Udenafil 150mg | Placebo
Number analyzed (Participants) | 141 | 140 | 147 | 141
Units on a Scale | 0.30 [0.04 to 0.57] | 0.65 [0.38 to 0.92] | 0.65 [0.39 to 0.91] | -0.06 [-0.32 to 0.21]
Statistical Analysis 1: Comparison: Udenafil 50 mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0566, ANCOVA; P-values are obtained from ANCOVA model with Baseline domain score and pooled site as covariates; Difference in LS Means = 0.36, 95% CI 2-sided [-0.01 to 0.73]
Statistical Analysis 2: Comparison: Udenafil 100 mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0002, ANCOVA; P-values obtained from ANCOVA model with Baseline domain score and pooled site as covariates; Difference in LS Means = 0.71, 95% CI 2-sided [0.34 to 1.08]
Statistical Analysis 3: Comparison: Udenafil 150mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0001, ANCOVA; P-values obtained from ANCOVA model with Baseline domain score and pooled site as covariates; Difference in LS Means = 0.71, 95% CI 2-sided [0.34 to 1.07]

7. Secondary Outcome: Change in Overall Satisfaction Domain Score Assessed by IIEF, Baseline to Week 12/Final Visit, mITT, LOCF
Description: Overall Satisfaction domain: 1/poor - 5/good scoring scale for each of 2 questions (2-10/good). Over last month, how satisfied have you been with your overall sex life? How satisfied have you been with your sexual relationship with your partner?
Time Frame: Baseline and Week 12
Population: mITT, LOCF
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a Scale
Arm/Group | Udenafil 50 mg | Udenafil 100 mg | Udenafil 150mg | Placebo
Number analyzed (Participants) | 141 | 140 | 147 | 141
Units on a Scale | 1.46 [1.07 to 1.85] | 2.15 [1.76 to 2.55] | 2.69 [2.31 to 3.07] | 0.60 [0.21 to 0.99]
Statistical Analysis 1: Comparison: Udenafil 50 mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0019, ANCOVA; P-values are obtained from ANCOVA model with Baseline domain score and pooled site as covariates; Difference in LS Means = 0.86, 95% CI 2-sided [0.32 to 1.40]
Statistical Analysis 2: Comparison: Udenafil 100 mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA; P-values are obtained from ANCOVA model with Baseline domain score and pooled site as covariates; Difference in LS Means = 1.55, 95% CI 2-sided [1.01 to 2.09]
Statistical Analysis 3: Comparison: Udenafil 150mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA; P-values are obtained from ANCOVA model with Baseline domain score and pooled site as covariates; Difference in LS Means = 2.09, 95% CI 2-sided [1.55 to 2.62]

8. Secondary Outcome: Global Assessment Questionnaire (GAQ), Week 12/Final Visit, mITT Population
Description: While Using the Study Medication, Did You Feel That Your Erections Improved (Yes Responders)
Time Frame: Week 12
Population: mITT
Measure: Number; unit: Yes Responders
Arm/Group | Udenafil 50 mg | Udenafil 100 mg | Udenafil 150mg | Placebo
Number analyzed (Participants) | 141 | 140 | 147 | 141
Yes Responders | 68 | 85 | 105 | 33
Statistical Analysis 1: Comparison: Udenafil 50 mg vs Udenafil 100 mg vs Udenafil 150mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Cochran-Armitage test
Statistical Analysis 2: Comparison: Udenafil 50 mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Chi-squared
Statistical Analysis 3: Comparison: Udenafil 100 mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Chi-squared
Statistical Analysis 4: Comparison: Udenafil 150mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Chi-squared

9. Secondary Outcome: Erectile Dysfunction Inventory of Treatment Satisfaction (EDITS) Derived Score, Subject Version, Week 12/Final Visit, LOCF, mITT
Description: EDITS -sum of responses (mapped to 0/bad-4/good scale, 11 questions standardized to scale of 100): How satisfied are you w/treatment? How likely to continue?, During past 4 wks, has treatment met expectations? How easy to use ? How satisfied w/how quickly it works? How long it lasts? How confident has it made you feel about ability to engage in sex? How satisfied is partner is with treatment effects? How does your partner feel about continuing use? How natural did process of achieving erection feel? Compared to before erection problem, how natural did erection feel in terms of hardness?
Time Frame: Baseline and Week 12
Population: mITT, LOCF
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a Scale
Arm/Group | Udenafil 50 mg | Udenafil 100 mg | Udenafil 150mg | Placebo
Number analyzed (Participants) | 141 | 140 | 147 | 141
Units on a Scale | 57.20 [53.13 to 61.27] | 64.16 [60.05 to 68.27] | 71.56 [67.59 to 75.53] | 44.55 [40.49 to 48.61]
Statistical Analysis 1: Comparison: Udenafil 50 mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANOVA; P-values are obtained from ANOVA model with pooled site as a covariate; Difference in LS Means = 12.65, 95% CI 2-sided [7.01 to 18.29]
Statistical Analysis 2: Comparison: Udenafil 100 mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANOVA; P-values are obtained from ANOVA model with pooled site as a covariate; Difference in LS Means = 19.61, 95% CI 2-sided [13.95 to 25.27]
Statistical Analysis 3: Comparison: Udenafil 150mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANOVA; P-values are obtained from ANOVA model with pooled site as a covariate; Difference in LS Means = 27.01, 95% CI 2-sided [21.44 to 32.59]

10. Secondary Outcome: Change From Baseline to Week 12/Final Visit in Mean Patient Self-Assessment of Erection (PSAE), mITT Population
Description: PASE: Chose one: 1) No evidence of tumescence or erection 2) partial tumescence or erection (not likely to be sufficient for penetration) 3) greater tumescence or erection sufficient for vaginal penetration, but not fully rigid 4) full rigidity; scale 1/poor, no evidence of erection - 4/good, full rigidity
Time Frame: Baseline and Week 12
Population: mITT
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a Scale
Arm/Group | Udenafil 50 mg | Udenafil 100 mg | Udenafil 150mg | Placebo
Number analyzed (Participants) | 141 | 140 | 147 | 141
Units on a Scale | 0.39 [0.29 to 0.49] | 0.49 [0.39 to 0.60] | 0.78 [0.69 to 0.88] | -0.05 [-0.15 to 0.05]
Statistical Analysis 1: Comparison: Udenafil 50 mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA; P-values are obtained from ANCOVA model with baseline PSAE score and pooled site as covariates; Difference in LS Means = 0.44, 95% CI 2-sided [0.30 to 0.57]
Statistical Analysis 2: Comparison: Udenafil 100 mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA; P-values are obtained from ANCOVA model with baseline PSAE score and pooled site as covariates; Difference in LS Means = 0.54, 95% CI 2-sided [0.40 to 0.68]
Statistical Analysis 3: Comparison: Udenafil 150mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA; P-values are obtained from ANCOVA model with baseline PSAE score and pooled site as covariates; Difference in LS Means = 0.83, 95% CI 2-sided [0.69 to 0.97]

11. Secondary Outcome: Change in SEP Question 1, Change From Baseline to Overall/Weeks 1-12, mITT
Description: SEP Question 1: Were you able to achieve at least some erection (some enlargement of the penis)? yes/no response. Percent yes responses at baseline compared with percent yes responses in overall study treatment period.
Time Frame: Baseline and Weeks 1-12
Population: mITT
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage Yes Responses
Arm/Group | Udenafil 50 mg | Udenafil 100 mg | Udenafil 150mg | Placebo
Number analyzed (Participants) | 141 | 140 | 147 | 141
Percentage Yes Responses | 3.39 [-0.18 to 6.97] | 3.16 [-0.44 to 6.75] | 9.28 [5.80 to 12.76] | -11.78 [-15.36 to -8.20]
Statistical Analysis 1: Comparison: Udenafil 50 mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA; P-values are obtained from ANCOVA model with proportion of "yes" responses during the baseline period and pooled site as covariates; Difference in LS Means = 15.18, 95% CI 2-sided [10.21 to 20.14]
Statistical Analysis 2: Comparison: Udenafil 100 mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 11, analysis 1]; Difference in LS Means = 14.94, 95% CI 2-sided [9.96 to 19.92]
Statistical Analysis 3: Comparison: Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 11, analysis 1]; Difference in LS Means = 21.06, 95% CI 2-sided [16.15 to 25.96]

12. Secondary Outcome: Change in SEP Question 4, Change From Baseline to Overall Study/Weeks 1-12, mITT
Description: SEP Question 4: Were you satisfied with the hardness of your erection? yes/no response. Percent yes responses at baseline compared with percent yes responses in overall study treatment period.
Time Frame: Baseline and Weeks 1-12
Population: mITT
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage Yes Responses
Arm/Group | Udenafil 50 mg | Udenafil 100 mg | Udenafil 150mg | Placebo
Number analyzed (Participants) | 141 | 140 | 147 | 141
Percentage Yes Responses | 27.12 [21.85 to 32.38] | 37.92 [32.63 to 43.21] | 43.42 [38.31 to 48.54] | 9.61 [4.35 to 14.86]
Statistical Analysis 1: Comparison: Udenafil 50 mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 11, analysis 1]; Difference in LS Means = 17.51, 95% CI 2-sided [10.22 to 24.81]
Statistical Analysis 2: Comparison: Udenafil 100 mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 11, analysis 1]; Difference in LS Means = 28.32, 95% CI 2-sided [21.01 to 35.62]
Statistical Analysis 3: Comparison: Udenafil 150mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 11, analysis 1]; Difference in LS Means = 33.82, 95% CI 2-sided [26.61 to 41.02]

13. Secondary Outcome: Change in SEP Question 5, Change From Baseline to Overall/Weeks 1-12, mITT
Description: SEP Question 5: Were you satisfied with this overall sexual experience? yes/no response. Percent yes responses at baseline compared with percent yes responses in overall study treatment period.
Time Frame: Baseline and Weeks 1-12
Population: mITT
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage Yes Responses
Arm/Group | Udenafil 50 mg | Udenafil 100 mg | Udenafil 150mg | Placebo
Number analyzed (Participants) | 141 | 140 | 147 | 141
Percentage Yes Responses | 26.27 [20.86 to 31.68] | 36.93 [31.48 to 42.38] | 41.88 [36.62 to 47.14] | 7.53 [2.13 to 12.94]
Statistical Analysis 1: Comparison: Udenafil 50 mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 11, analysis 1]; Difference in LS Means = 18.73, 95% CI 2-sided [11.23 to 26.23]
Statistical Analysis 2: Comparison: Udenafil 100 mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 11, analysis 1]; Difference in LS Means = 29.39, 95% CI 2-sided [21.86 to 36.92]
Statistical Analysis 3: Comparison: Udenafil 150mg vs Placebo; 540 subjects were randomized with 1:1:1:1 randomization scheme to the 4 treatment groups (placebo and udenafil 50mg, 100mg or 150mg). 135 subjects for each group vs. Placebo will provide at least 90% power with effect size from 0.41-0.44, 0.74-0.90 and 0.46-0.95 on 50 mg, 100 mg and 150 mg groups, respectively. Adjusted power is at least 90% using Bonferroni adjustment on hierarchical testing procedure. Considerations are based on results from Phase 2, Dong-A Study DA 2005-001(NCT00282607); Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 11, analysis 1]; Difference in LS Means = 34.35, 95% CI 2-sided [26.94 to 41.75]

ADVERSE EVENTS:
Time Frame: Twelve weeks
Arm/Group | Udenafil 50 mg | Udenafil 100 mg | Udenafil 150mg | Placebo
Serious Adverse Events (participants affected / at risk) | 1/147 | 1/148 | 3/154 | 1/150
Other Adverse Events (participants affected / at risk) | 43/147 | 51/148 | 49/150 | 11/150
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Udenafil 50 mg (N=147) | Udenafil 100 mg (N=148) | Udenafil 150mg (N=154) | Placebo (N=150)
Coronary Artery Stenosis (Cardiac disorders) | 0 | 0 | 0 | 1
Endocarditis (Infections and infestations) | 1 | 0 | 0 | 0
Small Intestinal Obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Angina Unstable (Cardiac disorders) | 0 | 0 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Lung Squamous Cell Carcinoma Stage Unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Udenafil 50 mg (N=147) | Udenafil 100 mg (N=148) | Udenafil 150mg (N=150) | Placebo (N=150)
Upper Respiratory Tract Infection (Infections and infestations) | 7 | 7 | 6 | 0
Nasopharyngitis (Infections and infestations) | 6 | 2 | 5 | 5
Sinusitis (Infections and infestations) | 2 | 4 | 2 | 2
Dyspepsia (Gastrointestinal disorders) | 1 | 7 | 4 | 0
Headache (Nervous system disorders) | 4 | 10 | 15 | 0
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 7 | 6 | 4 | 2
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 3 | 0
Flushing (Vascular disorders) | 9 | 8 | 10 | 0
Blood Creatine Phosphokinase Increased (Investigations) | 3 | 4 | 0 | 1
Blood Pressure Increased (Investigations) | 3 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less